CLINICAL TRIAL: NCT03335579
Title: Relationship Between General Anesthetic Mode and Postoperative Severe Cardiovascular and Cerebrovascular Complications: a Retrospective Cohort Study
Brief Title: General Anesthetic Mode and Postoperative Complications
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yan Zhou, MD, Principal Investigator, Peking University First Hospital
Other Study IDs: GATCIMACE
Record Dates: First submitted 2017-10-30; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Anesthesia
MeSH Terms: interventions — Inhalation; Anesthesia, General; Remifentanil; Sufentanil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-MACE: patients without major postoperative cardiac or cerebral complications
  Interventions: Combination Product: inhalation or propofol ,epidural or general anesthesia, remifentanil or sufentanil
- MACE: patients with major postoperative cardiac or cerebral complications
  Interventions: Combination Product: inhalation or propofol ,epidural or general anesthesia, remifentanil or sufentanil

INTERVENTIONS:
Combination Product: inhalation or propofol ,epidural or general anesthesia, remifentanil or sufentanil — Different combination of opioids and anesthetics

SUMMARY:
The relationship between anesthetic medication and postoperative major cardiac and cerebral complications will be studied using logistic regression model.

DETAILED DESCRIPTION:
The study group try to find out if there is a connection between the use of different anesthetic methods with different narcotic drugs and postoperative major cardiac and cerebral complications.

ELIGIBILITY:
Inclusion Criteria:

* non-cardiac surgery, with age> = 18 years old, ASA grade I-IV, under general anesthesia

Exclusion Criteria:

* non-general anesthesia, without the use of target-controlled infusion of remifentanil or sufentanil, absence of intraoperative or perioperative information.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients for non-cardiac surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 2016-12-31 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Major cardiac complication | 90 days after surgery
  major cardiac event

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Herling SF, Dreijer B, Wrist Lam G, Thomsen T, Moller AM. Total intravenous anaesthesia versus inhalational anaesthesia for adults undergoing transabdominal robotic assisted laparoscopic surgery. Cochrane Database Syst Rev. 2017 Apr 4;4(4):CD011387. doi: 10.1002/14651858.CD011387.pub2. PMID 28374886
- [Background] Flier S, Post J, Concepcion AN, Kappen TH, Kalkman CJ, Buhre WF. Influence of propofol-opioid vs isoflurane-opioid anaesthesia on postoperative troponin release in patients undergoing coronary artery bypass grafting. Br J Anaesth. 2010 Aug;105(2):122-30. doi: 10.1093/bja/aeq111. Epub 2010 Jun 23. PMID 20573633
- [Background] Min JJ, Kim G, Lee JH, Hong KY, Kim WS, Lee YT. Does the Type of Anesthetic Technique Affect In-Hospital and One-Year Outcomes after Off-Pump Coronary Arterial Bypass Surgery? PLoS One. 2016 Apr 7;11(4):e0152060. doi: 10.1371/journal.pone.0152060. eCollection 2016. PMID 27054364
- [Background] Guclu CY, Unver S, Aydinli B, Kazanci D, Dilber E, Ozgok A. The effect of sevoflurane vs. TIVA on cerebral oxygen saturation during cardiopulmonary bypass--randomized trial. Adv Clin Exp Med. 2014 Nov-Dec;23(6):919-24. doi: 10.17219/acem/37339. PMID 25618118